CLINICAL TRIAL: NCT04178421
Title: Computerized Eye-tracking Attention Training for Children With Special Needs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Chan Sui-yin Agnes, Professor Chan Sui-yin Agnes, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0298
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: ADHD; ASD; Learning Disorders
Keywords: Sustained attention; Impulse control; Eye-tracking; Special needs; Computerized training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Learning Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): A computerized eye -tracking program training the eye gaze fixation with the target to improve impulse control and sustained attention of children with special needs
  Interventions: Other: Computerized training program
- Control Group (Placebo Comparator): Computerized program
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Computerized training program — Eye-gaze fixation computer based training program
  Arms: Experimental Group
Other: Placebo — Pac-Man, Zookeeper, Tetris
  Other Names: Computerized program
  Arms: Control Group

SUMMARY:
Children with special needs (e.g. autistic spectrum disorder, attention deficit hyperactivity disorder) are found to have sustained attention problems. Several behavioral interventions have been carried out in the past to improve this situation. However, these interventions are often involved a high administration cost. Recently, researchers have been focusing on training the eye gaze fixation using the eye-tracking training games, as some of the research studies reported a correlation between atypical eye gaze patterns with poor sustained attention. The objective of the present study is to evaluate the effectiveness of a computerized eye-tracking attention training. Two batches of 48 primary school students will be recruited from email and the subject pool of the Department of Psychology of The Chinese University of Hong Kong. Participants are dividedly randomly and equally into either intervention or control group. Participants in both groups will undergo pre- and post-assessments measuring the executive function and attention before and after the intervention, respectively. However, there will be eight eye-tracking training sessions for the intervention group, but only the assessments are received in the control group. It is hypothesized that after the training, the performance of the training games and assessments will improve, indicated by increasing accuracy rates, as well as the reaction time of the tasks. The results would provide important information on the value of computerized eye gaze training and would guide the direction of interventions that target on improving the sustained attention and impulse control of children with special needs.

ELIGIBILITY:
Inclusion Criteria:

* a total of 96 primary school children (aged between 6 to 12 years) with special needs, defined by psychological disorders such as ASD, ADHD, ADD, and Dyslexia

Exclusion Criteria:

* Children with mental retardation will be excluded

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Flanker Inhibitory Control and Attention Test (Cognitive Test) | through study completion, an average of 2 year
  flanker inhibitory control and attention test to assess their attention
Dimensional Change Card Sort Test (Psychological Test Battery) | through study completion, an average of 2 year
  the Dimensional Change Card Sort Test to measure executive function

CONTACTS AND LOCATIONS:
Locations (1):
- Neuropsychology Laboratory, Department of Psychology, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided